CLINICAL TRIAL: NCT00937066
Title: Management of Patients With Moderate to Severe Asthma Uncontrolled When Treated With Low Dose Inhaled Corticosteroids: Cost-effectiveness of Three Therapeutics Alternatives
Brief Title: Cost-effectiveness Study of Symbicort as Maintenance and Reliever Therapy (SMART)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-RC0-SYM-2007/1
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
Keywords: Cost-effectiveness analysis; Symbicort
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Adult patients 18-65 years with moderate to severe uncontrolled asthma

SUMMARY:
This study is an economic evaluation of Symbicort (Budesonide/formoterol) as maintenance and reliever therapy (SMART) versus its competitive alternatives.

The aims of this study are:

* To estimate the relative effectiveness of each one of the alternatives in the management of patients with moderate to severe asthma through a systematic review for the following outcomes:

  * Cumulative incidence of asthma severe exacerbations symptoms
  * Safety of each alternative (frequency of adverse events and complications due to the medications)
* To estimate the direct medical costs of treating with each pharmacologic alternative: Symbicort as SMART versus increased use of inhaled corticosteroids or Adding long-acting inhaled beta 2 agonist plus inhaled corticosteroids.
* To create a decision analysis model (decision tree) that allows comparisons between the alternatives on expected values and costs.
* To calculate the average and incremental cost-effectiveness ratios.
* To carry out a sensitivity analysis to test de robustness of the cost-effectiveness results allowing for reasonable changes in expected values and costs.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe asthma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)

PRIMARY OUTCOMES:
Estimate incremental cost-effectiveness ratio using Symbicort as Maintenance and Reliever Therapy in the pharmacologic management of patients when compared with competitive alternatives | 12 months
Incremental cost-effectiveness ratio from using Symbicort as symbicort as Maintenance and Reliever Therapy when compared with its competitive alternatives | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Dennis, M.D., Study Director — Pontificia Universidad Javeriana; MARÍA XIMENA ROJAS, M.D., Principal Investigator — Pontificia Universidad Javeriana
Locations (1):
- Research Site, Bogotá, Colombia